CLINICAL TRIAL: NCT02497586
Title: Feasibility of Magnetic Resonance Spectroscopy in Lung Cancer
Acronym: MRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GN15ON255
Record Dates: First submitted 2015-06-15; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRS (Experimental): Magnetic resonance spectroscopy (MRS) is a type of scan which offers the possibility of assessing tumour function by measuring concentrations of chemicals (metabolites) within the abnormal tissue. This is a prospective feasibility study, aiming to recruit 15 consecutive patients with lung cancer to undergo proton MRS. The feasibility and repeatability of the technique will be assessed by analysis of the MR spectra obtained.
  Interventions: Radiation: Magnetic resonance spectroscopy

INTERVENTIONS:
Radiation: Magnetic resonance spectroscopy — Magnetic resonance spectroscopy (MRS) is a type of scan which offers the possibility of assessing tumour function by measuring concentrations of chemicals (metabolites) within the abnormal tissue. It is a well-established technique in imaging brain cancers.

SUMMARY:
Lung cancer is commonly characterised either with a surgical procedure or by taking a tissue sample with a needle. Unfortunately, these invasive approaches may be unsafe in many patients with lung cancer, who often have co-existing illnesses such as emphysema.

Magnetic resonance spectroscopy (MRS) is a type of scan which offers the possibility of assessing tumour function by measuring concentrations of chemicals (metabolites) within the abnormal tissue. It is a well-established technique in imaging brain cancers. It has also been more recently studied in assessing prostate, liver and heart. There has been very little exploration of the potential role of MRS in lung cancer.

The proposed feasibility study will recruit 15 patients with proven lung cancer to undergo an MRS scan. The reliability of the technique for metabolite measurement will be determined by comparing repeated scans from the same region in the same tumour. Further scans from different regions in the same tumour, normal lung around the tumour and tumour regions in different patients will be used to look for any patterns in the cancer metabolites which may indicate avenues for potential future research.

DETAILED DESCRIPTION:
Magnetic resonance spectroscopy (MRS) is a magnetic resonance imaging (MRI) application that we aim to utilise in lung cancer for the first time at a higher magnetic field strength (3 Tesla). MRS allows nuclear magnetic resonance spectra to be obtained from user-defined regions of interest (ROIs) within body tissues. These spectra can be used to quantify concentrations of tumour metabolites, providing unique biological information non-invasively and without the need for ionising radiation or intravenous contrast material. Proton MRS is a well-established technique for characterisation of brain pathology and prostate cancer. MRS in the lung is more challenging as it is a moving structure but has been shown to be feasible in a previous small study using more basic standard field strength equipment and technique. MRS of other moving structures, namely the heart and liver, has been shown to be achievable.

It is believed that MRS, using a higher field strength (3 Tesla) machine, has not been applied before in the evaluation of lung cancer in human subjects. Successful utilisation of this technology to quantify metabolite concentrations within lung cancers offers new opportunities for non-invasive tumour classification. For example, low tumour oxygen levels, a known prognostic indicator, may be identifiable by non-invasive measurement of lactate concentration by MRS. Since MRS is an easily repeatable technique without ionising radiation, it may also prove useful in response assessment following lung cancer therapies. This is a prospective feasibility study, aiming to recruit 15 consecutive patients with lung cancer to undergo proton MRS. The feasibility and repeatability of the technique will be assessed by analysis of the MR spectra obtained.

The principal research questions is: Can MRS scans be obtained in lung cancer with a high field strength (3 Tesla) MR scanner? The secondary research questions are: Is there any indication of reproducibility in the MRS signals obtained? Is there any indication of MRS patterns correlating with tumour type and other clinical parameters which might be a useful subject for further investigation in lung cancer characterisation?

Summary of interventions:

1. During attendance at respiratory clinic, invite patient to participate in study and issue Patient Information Sheet (PIS), highlighting contact details for next steps (typically 5 min)
2. Patients with questions may contact a study investigator using the telephone number in the PIS to have them answered (typically 5-15 min)
3. Patients wishing to proceed contact the RIF using the telephone number in the PIS to arrange a convenient scan appointment and taxi transfers (typically 5 min) At least 1 day after clinic attendance
4. Written informed consent obtained, pre-scan checklist completed and GP letter sent by medical member of study team. Research radiographer completes safety checklist with patient. Scan undertaken, with maximum 'on table' scan time of 1 hour.

Implications for research for future service developments:

If this early study shows MRS of lung cancer to be technically feasible, the investigators will apply for external funding for a larger prospective study or studies correlating the MRS findings with a panel of clinical, imaging, histopathological and molecular variables. These secondary studies would have potential to alter clinical practice in tumour characterisation and follow-up. The overall aim of the research would be the development of a non-invasive tool to enable diagnosis and characterisation of suspected lung cancers.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-confirmed small cell or non-small cell lung cancer
* solid intrapulmonary tumour of at least 3 cm in long and short axis diameters on transverse CT images
* ECOG performance status ≤ 2
* able to provide written informed consent and respond appropriately to verbal instructions for scan acquisition
* age 18 years or older

Exclusion Criteria:

* chemotherapy within the preceding 12 months
* previous radiotherapy to the tumour
* cardiac pacemaker/defibrillator, internal pacing wires, cerebral aneurysm clip, incompatible metallic heart valve replacements, other incompatible implants/prostheses, claustrophobia or other MRI contraindication
* history of metal entering the body or eye, unless residual metal in the affected area likely to cause harm has been adequately excluded by X-ray in the opinion of Dr Cowell or Dr Stobo
* intractable cough, inability to lie flat or other impediment to acquisition of breath-held MR images
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Presence of metabolite peaks | Data collected on day 1
  Presence of metabolite peaks in MR spectra obtained from lung tumours using a 3T MR system.

SECONDARY OUTCOMES:
Reproducability of metabolite peaks | Data collected on day 1
  Reproducibility of metabolite peak ratios in MR spectra repeatedly obtained from lung tumours using a 3T MR system.
Metabolite peak-clinical parameter colleration | Data collected on day 1
  Correlation between metabolite peak ratios in MR spectra from lung tumours and clinical parameters including lung cancer type and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: David B Stobo, Dr, Principal Investigator — NHS Greater Glasgow and Clyde

REFERENCES:
- [Background] Castillo M, Kwock L, Mukherji SK. Clinical applications of proton MR spectroscopy. AJNR Am J Neuroradiol. 1996 Jan;17(1):1-15. No abstract available. PMID 8770242